CLINICAL TRIAL: NCT02252796
Title: Phase I Dose Escalation Study of a Hypofractionated Stereotactic Boost (HySBst) to the Primary Site in Patients With Stage II-III Non-small Cell Lung Cancer
Brief Title: Phase I Hypofractionated Stereotactic Boost (Radiotherapy) for Non-Small Cell Lung Cancer
Acronym: HySBst
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WVU020513
Record Dates: First submitted 2014-09-25; First posted 2014-09-30 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Radiotherapy Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sub-group 1 (Experimental): HySBst to be delivered during week 1 with Chemo-radiation to be delivered weeks 2-7
  Interventions: Radiation: Hypofractionated Stereotactic Boost; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Image-guided IMRT
- Sub-group 2 (Experimental): Chemo-radiation to be delivered weeks 1-6 and HySBst to be delivered week 7
  Interventions: Radiation: Hypofractionated Stereotactic Boost; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Image-guided IMRT

INTERVENTIONS:
Radiation: Hypofractionated Stereotactic Boost — An ablative dose of radiation is delivered to the primary tumor target over a week through Stereotactic Ablative Radiotherapy.
  Other Names: HySBst
Drug: Carboplatin — Given during chemo-radiation phase and optional consolidative phase.
Drug: Paclitaxel — Given during chemo-radiation phase and optional consolidative phase.
Radiation: Image-guided IMRT — Given during chemo-radiation phase

SUMMARY:
This study will help researchers test the safety of hypofractionated dose of radiotherapy (HySBst) at different dose levels before or after chemo-radiation for Non Small Cell Lung Cancer.

DETAILED DESCRIPTION:
Patients are assigned to Sub-group 1 or 2 based on the primary lesion size and location. This protocol will utilize a standard 3 + 3 phase I design with three patients enrolled per cohort.

Patients will be offered the opportunity to participate in the blood specimen component of the study.

Patients will be followed up to 2 years post radiation therapy.

Sub-group 1 will receive HySBst for 1 week. Weeks 2-7 will be standard chemo-radiation therapy. Patients have the option of consolidative chemotherapy at week 12.

Sub-group 2 will receive standard chemo-radiation therapy for weeks 1-6 then receive HySBst during week 7. Patients have the option of consolidative chemotherapy at week 12.

HySBst dose escalation for each sub-group is listed below:

Optional: 4 Gy x 4 daily fractions Level 1: 5 Gy x 4 daily fractions Level 2: 5.5 Gy x 4 daily fractions Level 3: 6 Gy x 4 daily fractions

DLTs will be based on events occurring during the course of HySBst.

Chemo-Radiation Therapy is defined as:

Standard Carboplatin & Paclitaxel Doublelet Regimen with weekly Carboplatin AUC 2/week and Paclitaxel 45 mg/ m2/ week during conventionally fractionated IMRT

Image-guided IMRT to 60 Gy, 5 x per week for 6 weeks

Consolidative chemotherapy is defined as Carboplatin AUC 6 and Paclitaxel 200 mg/m2 every 21 days x 2 cycles will be given after ALL radiotherapy is delivered.

ELIGIBILITY:
Inclusion Criteria:

* Stage II - III Non Small Cell Lung Cancer

Exclusion Criteria:

* Primary tumor directly invading into any mediastinal structures, such as the heart, major blood vessels, esophagus, trachea, and the proximal bronchial tree.
* Prior chemotherapy for NSCLC
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
* Severe, active co-morbidity
* Pregnancy or women of childbearing potential
* Any history of allergic reaction to paclitaxel or other taxanes, or to carboplatin
* Uncontrolled neuropathy ≥ grade 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-07; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of HySBst | 2 years

SECONDARY OUTCOMES:
Dose Limiting Toxicity | 1 week
Blood Sample Collection | 2 years
  Biomarker analysis
Local Control | 2 years
  To determine the 2-year regional, and distant metastasis rates, progression-free survival (PFS), local progression free survival (L-PFS), overall survival (OS)
Quality of Life | 2 years
  To determine the quality of life before and after treatment using the European Organisation of Research and Treatment of Cancer Quality of Life Questionnaire, Core 30 and Lung Cancer 13 (EORTC QLQ-C30, and the LC 13) scales

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Mattes, MD, Principal Investigator — West Virginia University - Mary Babb Randolph Cancer Center
Locations (1):
- West Virginia University Hospitals Mary Babb Randolph Cancer Center, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No